CLINICAL TRIAL: NCT03400982
Title: Reference Curve on Bone Mineral Density in Men
Acronym: COURDO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2017-10
Record Dates: First submitted 2017-12-07; First posted 2018-01-17 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Bone Mineral Density; Grip Strength; Physical Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone Mineral Density (Experimental): Bone densitometry measurement: measurement of bone mineral densitometry with bone densitometry
  Interventions: Diagnostic Test: Bone densitometry measurement

INTERVENTIONS:
Diagnostic Test: Bone densitometry measurement — Bone densitometry and measurement of body composition

SUMMARY:
In men, the hope of lower life, the absence of equivalent of menopause and the existence of a higher peak bone mass are the three factors that explain the lower incidence of osteoporosis in men.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 20 and 30 years
* Caucasians

Exclusion Criteria:

* Lack of express consent
* Pieces of metal or plastic parts in field
* Diseases which cause technical difficulties for the correct evaluation of the hip and spine (severe dysplasia, hip surgery or lumbar spine)
* Adult protect buy the law

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Bone mineral density of the spine | Day 0
  to establish reference curves in elderly mal volunteers from 20 to 30 years through the assessment of bone mineral density of the spine
Bone mineral density of the hip | Day 0
  to establish reference curves in elderly mal volunteers from 20 to 30 years through the assessment of bone mineral density of the hip

SECONDARY OUTCOMES:
Fat mass of the body | day 0
  to establish reference curves in elderly mal volunteers from 20 to 30 years through the assessment of body composition
Lean mass of the body | day 0
  to establish reference curves in elderly mal volunteers from 20 to 30 years through the assessment of body composition

CONTACTS AND LOCATIONS:
Overall Officials: Eric LESPESSAILLES, Principal Investigator — CHR Orléans
Locations (3):
- France (3):
  - CHU Amiens, Amiens
  - Hopital Lariboisiere, Paris
  - CHU de Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrahamsen B, Hansen TB, Jensen LB, Hermann AP, Eiken P. Site of osteodensitometry in perimenopausal women: correlation and limits of agreement between anatomic regions. J Bone Miner Res. 1997 Sep;12(9):1471-9. doi: 10.1359/jbmr.1997.12.9.1471. PMID 9286764
- [Background] Smotherman MS, Narins PM. Effect of temperature on electrical resonance in leopard frog saccular hair cells. J Neurophysiol. 1998 Jan;79(1):312-21. doi: 10.1152/jn.1998.79.1.312. PMID 9425200
- [Background] Baumgartner RN. Body composition in elderly persons: a critical review of needs and methods. Prog Food Nutr Sci. 1993 Jul-Sep;17(3):223-60. PMID 8234779